CLINICAL TRIAL: NCT00434733
Title: A Phase III, Randomized, Controlled, Observer-Blind, Multicenter Study to Evaluate the Immunogenicity, Safety and Tolerability of Two Doses of FLUAD-H5N1 Influenza Vaccine in Adult and Elderly Subjects
Brief Title: Immunogenicity, Safety and Tolerability of Two Doses of FLUAD-H5N1 Influenza Vaccine in Adult and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V87P4; 2006-005428-18
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Influenza
Keywords: Influenza H5N1, pandemic
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Pandemic influenza vaccine

SUMMARY:
This study is designed to evaluate the immunogenicity, safety and tolerability of 2 doses of FLUAD-H5N1 vaccine compared to 2 doses of trivalent, interpandemic FLUAD, each administered 3 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects 18 years of age who signed the informed consent

Exclusion Criteria:

* Receipt of another investigational agent within 4 weeks
* Receipt of influenza vaccination for current season 2006/2007.
* any acute disease or infection, history of neurological symptoms or signs, known or suspected impairment of immune function, any serious disease, bleeding diathesis
* fever (defined as axillary temperature ³38.0°C) within 3 days (prior to Visit 1)
* Pregnant or breastfeeding or females of childbearing potential who refuse to use an acceptable method of birth control
* Surgery planned during the study period
* Hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the study vaccine
* Receipt of another vaccine within 3 weeks prior to Visit 1 or planned vaccination within 3 weeks following the last study vaccination
* History of (or current) drug or alcohol abuse
* Any condition, which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Adverse event rate

SECONDARY OUTCOMES:
Seroconversion and seroprotection after two doses of H5N1 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics GmbH & Co KG Novartis, Study Chair — Novartis Vaccines and Diagnostics GmbH & Co KG., Germany
Locations (1):
- Centrum Badań Farmakologii Klinicznej monipol, Krakow, Poland